CLINICAL TRIAL: NCT04515381
Title: Mardin Artuklu University Of Scientific Research Projects
Brief Title: Title: Effect of Therapeutic Touch on Daytime Sleepiness, Stress and Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Birgül Vural Doğru, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MAU.SRP.SH.005
Record Dates: First submitted 2020-08-06; First posted 2020-08-17 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Stress; Fatigue; Sleepiness
Keywords: Therapeutic touch; Daytime sleepiness; Sleep quality; Stress; Fatigue; Nurse-midwifery student
MeSH Terms: conditions — Fatigue; Sleepiness; Disorders of Excessive Somnolence; Sleep Initiation and Maintenance Disorders | interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic touch group (Experimental): Each student from the Therapeutic touch (TT) group was given TT sessions via Krieger-Kunz method in a total of 8 times in the manner of twice a week for one group (Monday - Wednesday) and another group (Tuesday - Thursday) for a duration of 1 month (4 week). TT application procedure: The procedure was explained to the student, the student person was concentrated, concentrated practitioner for TT application, the student's entire body was evaluated from head to foot with the practitioner's hands at a distance of about 2 inc, hands were moved regularly and rhythmically to prevent imbalances in the energy field, the energy field was re-evaluated from top to bottom and rebalanced if there was a blocked area, finally, the student was left to rest and response to the treatment was observed. The TT sessions of 20 minutes were applied on the students and they were given a short rest at the end of the session
  Interventions: Other: Therapeutic Touch
- Placebo group (Placebo Comparator): For students in the placebo group, the similar duration (20 minutes) and frequency (2 sessions a week, total of 8 sessions) of TT was applied with hands at a certain distance from the body (approximately 5 cm) and they were moved without a specific order. The application was performed by the other researcher in a separate room to the placebo group.
  Interventions: Other: Sham Therapeutic Touch
- Control group (Other): There was no attempt being made towards the students within the control group. At the end of the 4th week, all students were asked to repeat measurements
  Interventions: Other: Control group

INTERVENTIONS:
Other: Therapeutic Touch — Therapeutic Touch
  Arms: Therapeutic touch group
Other: Control group — Making measurements at the beginning of the research and 4 weeks
  Arms: Control group
Other: Sham Therapeutic Touch — Sham Therapeutic Touch
  Arms: Placebo group

SUMMARY:
Objective: This study was conducted to assess the effect of therapeutic touch on stress, daytime sleepiness, sleep quality and fatigue among the students of nursing and midwifery.

Design: Randomized placebo-controlled study.

DETAILED DESCRIPTION:
The trial was conducted between April and July 2018. The students who met the inclusion criteria were separated into three groups through randomization method as in therapeutic touch (n=32), placebo (n=32) and control (n=32), and a total of 96 students participated in the study. In this randomized placebo controlled study, the therapeutic touch group were subjected to therapeutic touch for twice a week throughout 4 weeks with each session of 20 minutes. The data was acquired via Student Information Form, Epworth Sleepiness Scale, Pittburgh Sleep Quality Index, Perceived Stress Scale and Visual Analogue Scale for Fatigue.

ELIGIBILITY:
Inclusion Criteria:

* students who were at and above the age of 18,
* were the 1st year, 2nd year, 3rd year or 4th year students of nursing or midwifery,
* did not receive any energy therapy (Reiki, healing touch, therapeutic touch),
* received a score above 10 from the Epworth sleepiness scale (ESS),
* did not have any communication problem,
* and accepted to take part in the study were included in the study.

Exclusion Criteria:

* Students who were getting a psychologic and/or pharmacologic treatment in regard to their sleep, fatigue and stress problems,
* previously got a psychiatric diagnosis, still had a psychiatric illness,
* previously or still used anxiety (psychotropic) medicines were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale | Change from baseline and 4 weeks.
  The score of PSS-10 varied from 0 to 40. High score shows the excessiveness of the perceived stress of the individual
Change in Epworth Sleepiness Scale | Change from baseline and 4 weeks.
  The scale consists of 8 items and score varies from 0-24. If the total score is between 2-10, it is considered as normal, pathological sleepiness indicator is greater than 10, thirteen and higher values are considered excessive daytime sleepiness.
Change in Pittsburgh Sleep Quality Index | Change from baseline and 4 weeks.
  In PSQI analysis, 18 items were scored and there are 7 categories as in subjective sleep quality, delayed sleep, sleep duration, accustomed sleep activity, sleep disorder, use of sleeping pill and daytime dysfunction. Total score varies from 0 to 21. If the total PSQI score is ≤5, it stands for "good sleep quality", and if the score is >5, it stands for "bad sleep quality"
Change in Visual Analogue Scale | Change from baseline and 4 weeks.
  The scale of fatigue is a scale of 10 cm that assesses the severity of the fatigue in the last week. The left side of the scale contains the label of "I do not feel fatigue", while the right side of the scale contains the label of "I Feel Extreme Fatigue and Exhaustion". VASF value is determined through the measurement of the distance between the very left side of the scale and the marked point

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No